CLINICAL TRIAL: NCT02489682
Title: Clinical Informed Consent Format Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: ICON plc (Industry)
Responsible Party: Principal Investigator, Tamar Krishnamurti, Research Scientist, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A016520
Record Dates: First submitted 2015-06-24; First posted 2015-07-03 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Consent Forms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Informed Consent Format - short written (Experimental): Intervention to be administered:
  - Short-form written informed consent information, followed immediately by outcomes questionnaire
  Interventions: Other: Short-form written Informed consent information
- Informed Consent Format - long written (Experimental): Intervention to be administered:
  - Long-form written informed consent information, followed immediately by outcomes questionnaire
  Interventions: Other: Long-form written Informed consent information
- Informed Consent Format - video (Experimental): Intervention to be administered:
  - Video informed consent information, followed immediately by outcomes questionnaire
  Interventions: Other: Video Informed consent information

INTERVENTIONS:
Other: Long-form written Informed consent information
  Arms: Informed Consent Format - long written
Other: Short-form written Informed consent information
  Arms: Informed Consent Format - short written
Other: Video Informed consent information
  Arms: Informed Consent Format - video

SUMMARY:
This study evaluates the effectiveness of a patient-centered short written informed consent form and a patient-centered short video informed consent in a randomized controlled trial (control = traditional informed consent ). Primary outcome measures include critical knowledge acquisition, risk and benefit judgments, and desired enrollment in a hypothetical clinical trial. The investigators hypothesized that the patient-centered patient-designed consent forms (video and written format) would do as well as or outperform the traditional consent form on the primary outcomes.

DETAILED DESCRIPTION:
Traditional informed consent documents tend to be lengthy and technical, often too dense to facilitate proper patient-engagement. In this study, the investigators test the effectiveness of a previously developed patient-centered, short informed consent document and a patient-centered, short informed animated consent video as compared to a lengthy traditional informed consent document for the same clinical condition (i.e. severe asthma)

In this study, self-identified asthma patients, aged 18 or older, attending an experimental session in a university computer laboratory will be randomly assigned to read either the full informed consent document (control) or the short, patient-centered informed consent document or to view the short patient-centered informed consent video. Participants will also complete a follow-up survey at 1-week.

The main outcome measures are:

Engagement in the information (1=not at all engaged, 2=not very engaged, 3= somewhat engaged, 4=very engaged, 5=completely engaged).

Intention to enroll in the clinical trial

(1=definitely would not, 3=neutral, and 5=definitely would)

Trial knowledge (12 multiple choice questions, e.g. ""When can [the participants] withdraw from the trial?")

Trust in the clinical trial physician (Six questions beginning with, "If [the participant] decided to enroll in this study, how much would [the participant] trust Dr. Janet Taylor, the physician who is leading the study, to...")

Perceived risks and benefits of the trial (Four questions, e.g. "Imagine that [the participant] enrolled in the clinical trial, how likely do [the participants] think it is that the drug would be more effective in treating [the participant's] asthma symptoms than an average asthma drug on the market?")

The investigators hypothesize that the two experimental conditions will outperform the control condition on engagement and trial knowledge and would do as well as the control on the remaining outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* fluent in English
* self-identifying as asthma patients

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Hypothetical trial enrollment as assessed by a likelihood of enrollment question | immediately after intervention
Engagement as assessed by a likert scale engagement question | immediately after intervention
Trust in physician as assessed by a composite of likert scale questions measuring trust | immediately after intervention
Trial Knowledge as assessed by a composite of 12 true/false questions | immediately after intervention
Perceived Risk and Benefit as assessed by a series of judgment questions | immediately after intervention

SECONDARY OUTCOMES:
Change in hypothetical trial enrollment as assessed by a likelihood of enrollment question at 1 week from intervention | 1-week follow-up
Change in trust in physician as assessed by a composite of likert scale questions measuring trust at 1 week from intervention | 1-week follow-up
Change in hypothetical trial trial knowledge as assessed by a composite of 12 true/false questions at 1 week from intervention | 1-week follow-up
Change in Perceived Risk and Benefit as assessed by a series of judgment questions at 1 week from intervention | 1-week follow-up